CLINICAL TRIAL: NCT05580068
Title: Pilot-Studie Zur Explorativen Untersuchung Und Validierung Eines Studienvorhabens Zur Digitalen Therapiesteuerung Von Patienten Mit Arterieller Hypertonie im Vergleich Der Behandlung Mit Dem Standard-of-Care - iATROS eXPLORE
Brief Title: Investigation and Validation of a Study Project on Digital Therapy Management of Patients With Arterial Hypertension
Acronym: eXPLORE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: iATROS GmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 02
Record Dates: First submitted 2022-10-11; First posted 2022-10-14 (Actual); Last update posted 2024-03-06 (Actual); Status verified 2024-03

CONDITIONS: Cardiovascular Diseases; Hypertension
Keywords: eHealth; cardiology; hypertension
MeSH Terms: conditions — Cardiovascular Diseases; Hypertension

STUDY DESIGN:
Intervention Model Description: monocentric randomized controlled study (RCT)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): The intervention to be carried out in the treatment group is the use of the therapy measures for the treatment of arterial hypertension, which is delivered through the iATROS medical device. The therapy by means of the medical device takes place over 90 days.
  Interventions: Device: Hypertension therapy through iATROS medical device
- Control Group (No Intervention): For the duration of the in-life phase, the treatment of the control group will follow the standard-of-care except for the measures necessary for the conduct of the study.

INTERVENTIONS:
Device: Hypertension therapy through iATROS medical device — The intervention to be carried out in the treatment group is the use of the therapy support provided by the iATROS medical device for the treatment of arterial hypertension.
  In particular, patients are guided through a structured digital therapy program that enables them to better manage their disease. Patient receive reminders for taking their medication, for performing vital parameter measurements, and receive educational content for them to learn how to manage their disease better.
  Arms: Intervention Group

SUMMARY:
The purpose of this pilot study is to exploratively test the basic feasibility of a clinical trial for the controlled investigation of the efficacy and effectiveness of iATROS digital therapy management in the treatment of patients with arterial hypertension within the framework of a clinical trial. In addition, the results of the treatment will be used to generate an initial data basis for the effectiveness of treatment with iATROS.

DETAILED DESCRIPTION:
The aim of this pilot project is to form the basis for testing the iATROS platform in an controlled setting of a clinical study, in particular to collect data for a more precise determination of the sample size including the investigation of dropout rates, to investigate the acceptance of study-related measures, and to test and better prepare the procedures for the successful implementation of study-related measures. Furthermore, the first data for testing the effectiveness of the iATROS solution for the treatment of hypertensive patients will be collected. For this purpose, health data as well as data points on health literacy and patient sovereignty will be collected from the patients in the pilot study.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 18 years of age
* Existing diagnosis of arterial hypertension according to ICD-10 I10.- to I13.-, i.e. presence of the disease is recorded at the time of inclusion in the study.
* Blood pressure at the time of inclusion is ≥130 mmHg systolic (24h mean) at 24h blood pressure measurement or, alternatively, at-home blood pressure measurement at ≥135 mmHg systolic (mean of 7 days). In case of the presence of a 24-h blood pressure measurement, this value is decisive compared to the at-home measurement.
* Possession and use of a smartphone that allows the installation and use of "iATROS", whereby "use" implies that the patient possesses the physical and mental abilities to use and apply the iATROS app

Exclusion Criteria:

* Lack of capacity to consent
* < 18 years of age
* No use of a smartphone
* Lack of the physical and mental abilities necessary to use the iATROS app, or generally to use so-called "apps" on a smartphone or tablet.
* Tumor disease associated with a reduced life expectancy of less than 1 year
* Immunosuppression
* Advanced dementia
* Any other disease associated with a reduced life expectancy of less than 1 year
* Any disease/condition that limits participation in the program
* Pregnant or breastfeeding patients
* A secondary hypertension known to the patient (by history)
* Blood pressure at inclusion is >170mmHg systolic on 24h blood pressure measurement (24h mean) or, alternatively, the at-home blood pressure measurement is >175mmHg systolic (mean value of the 7 days). In case of a 24h blood pressure measurement, this value is decisive compared to the at-home measurement.
* Existing participation and enrollment in the iATROS hypertension health program.
* Participation in another clinical trial, if complications with compliance, the measures to be performed, a distortion of the results, or the status of a treatment according to the current standard of care result from the participation.
* Comorbidities or the presence of any other physical condition that would prohibit the use of the ESC Hypertension Guideline of 2018 as target blood pressure (i.e. if, due to the patient's individual situation, a different value should be given as a target value for a blood pressure value to be classified as healthy).
* Addictions
* Stroke in the last 3 months
* Transient ischemic attack (TIA) in the last 3 months

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2022-11-10 (Actual); Primary Completion 2024-10 (Estimated); Study Completion 2024-10 (Estimated)

PRIMARY OUTCOMES:
Exploratory testing of study-related measures and the use of iATROS. | Baseline and study completion, an average of 180 days
  Determination of subjective burden perception of the study-related measures using the Study Participant Feedback Questionnaire (SPFQ) - Questionnaire.
  The three subscales (A-C) are administered at three discrete time points, immediately after enrolment, after half the in-live phase time has passed and at the last visit in the study center. The questions are answered on a 5-point scale with a higher level indicating a higher satisfaction with the study-related measures. Possible levels are 0 to 24 (subscale A), 0 to 39 (subscale B) and 0 to 14 (subscale C).

SECONDARY OUTCOMES:
Blood pressure reduction | Baseline and 90 days after enrolment
  Measurement of blood pressure in mmHg after 90 days of treatment as compared to baseline.
  Comparison of the mean absolute reduction in systolic blood pressure in intragroup analysis per study arm and between treatment arms (intervention vs. control).
Blood pressure classification | Baseline, 90 days, and 180 days after enrolment
  Assessment of the fraction of patients in [%] with a blood pressure classified as "healthy" as per the definition outlined in the "2018 ESC/ESH Clinical Practice Guidelines for the Management of Arterial Hypertension " after 90 days of treatment and at follow-up at 180 days as compared to baseline. Comparison of the mean absolute reduction in systolic blood pressure in intragroup analysis per study arm and between treatment arms (intervention vs. control).
Health Literacy Questionnaire (HLQ) | Baseline and 90 days after enrolment
  Administration of the Health Literacy Questionnaire (HLQ) to assess disease-related health literacy.
  The questionnaire is comprised of 9 subscales. Scale 1-5 are graded on a 4-point scale (possible levels per subscale 1 to 4), scale 6-9 are graded on a 5-point scale (possible levels per subscale 1 to 5) with higher levels showing higher health literacy.
  Measurement at baseline and at the end of a 90-day treatment period. Assessment of changes in health literacy in intra-group comparison per study arm and inter-group comparison.
Patient Activation Measure (PAM) | Baseline and 90 days after enrolment
  Measurement of degree of patient activation via the Patient Activation Measure (PAM) questionnaire.
  Measurement at baseline and at the end of a 90-day treatment period. Assessment of changes in health literacy in intra-group comparison per study arm and inter-group comparison.
  Possible levels 0 to 100, with a higher level indicating higher activation.
Blood pressure reduction effect stability | 90 days and 180 days after enrolment
  Measurement of blood pressure level in mmHg 90 days after finishing in-live phase and comparison to blood pressure level 90 days after enrolment.
  Comparison of the mean absolute reduction in systolic blood pressure in intragroup analysis per study arm and between treatment arms (intervention vs. control).

CONTACTS AND LOCATIONS:
Overall Officials: Stefan Brunner, Prof. Dr., Principal Investigator — Medizinische Klinik und Poliklinik 1, Ludwig-Maximilians-University of Munich
Locations (1):
- Medizinische Klinik und Poliklinik 1, Ludwig-Maximilians-University of Munich, Munich, Bavaria, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Schlichtiger J, Struven A, Massberg S, von Degenfeld G, Leber A, Weyh P, Meyer J, Brunner S, Stremmel C. Evaluation of a digital therapy programme for the treatment of primary arterial hypertension: eXPLORE - study protocol for a fully decentralised randomised controlled feasibility study. BMJ Open. 2024 Sep 5;14(9):e081347. doi: 10.1136/bmjopen-2023-081347. PMID 39237273